CLINICAL TRIAL: NCT02234999
Title: A Phase 1, Single-center, Open-label Study to Evaluate the Metabolism and Excretion of [14C]-CC-122 in Healthy Male Subjects
Brief Title: Radiolabeled Study of CC-122 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: CC-122-CP-003
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics, Healthy Subjects
MeSH Terms: interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3mg [14C]-CC-122 (Single Dose) (Experimental): Single oral capsule of 3mg [14C]-CC-122. given as a suspension under fasting conditions on Day 1
  Interventions: Drug: CC-122

INTERVENTIONS:
Drug: CC-122 — 3mg [14C]-CC-122 will be administered as a single dose

SUMMARY:
To evaluate the metabolism and excretion of [14C]-CC-122 in healthy male subjects

DETAILED DESCRIPTION:
This is a single-center, open-label study to evaluate the metabolism and excretion of [14C]-CC-122 following a single oral dose of [14C]-CC-122 in healthy male subjects. It is planned for 6 subjects to be enrolled; each subject will participate in a screening phase, a baseline phase, a treatment phase, and a follow up phone call. Blood, urine and fecal samples will be collected for analyses.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy adult male of any race and between 18 years of age to 55 years of age, inclusive, at the time of signing the informed consent document.

  2. Understand and voluntarily sign an informed consent document before any study related assessments/procedures are performed.

  3. Able to adhere to the study visit schedule and other protocol requirements. 4. Must practice true abstinence or agree to use a condom (a latex condom is recommended) during sexual contact with a pregnant female or a female of childbearing potential while participating in the study and for at least 28 days following discontinuation of investigational product, even if he has undergone a successful vasectomy.

  5. Must agree to abide by the CC 122 Pregnancy Prevention Risk Management Plan 6. Must have a body mass index between 18 and 33 kg/m2, inclusive, at screening.

  7. Must be healthy as determined by the Investigator on the basis of medical history, physical exam, clinical laboratory test results, vital signs, and 12-lead electrocardiogram at screening:
  * Must be afebrile (febrile is defined as ≥ 38.5°C or 101.3°F)
  * Supine systolic blood pressure must be in the range of 90 to 140 mmHg, supine diastolic blood pressure must be in the range of 50 to 90 mmHg, and pulse rate must be in the range of 40 to 110 bpm
  * Normal or clinically acceptable 12 lead electrocardiogram, with a QTcF value ≤ 430 msec

Exclusion Criteria:

* 1. History of any clinically significant and relevant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies (including a known hypersensitivity to a member of the class of IMiDs®), or other major disorders.

  2. Any condition, including the presence of clinically significant laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study.

  3. Any condition that confounds the ability to interpret data from the study. 4. Exposed to an investigational drug (new chemical entity) within 30 days preceding dose administration, or five half lives of that investigational drug, if known (whichever is longer).

  5. Participation in more than one other radiolabeled investigational drug study within 12 months prior to check in.

Note: The previous radiolabeled investigational drug must have been received more than 6 months prior to check in and the total planned exposure from this current study and the previous study must be within the recommended levels considered safe, per United States Code of Federal Regulations governing Protection of Human Subjects; radioactive drugs for certain research uses.

6. Exposure to significant radiation (for example, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to check in.

7. Used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days of dose administration.

8. Used any nonprescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of dose administration.

9. Used cytochrome P450 3A inducers and/or inhibitors (including St. John's wort) within 30 days of dose administration.

10. Received a live vaccination within 90 days of dose administration. 11. Has any surgical or medical conditions possibly affecting absorption, distribution, metabolism, and/or elimination, for example, bariatric procedure, or plans to have elective or medical procedures performed during the conduct of the trial. Prior appendectomy is acceptable, but prior cholecystectomy would result in exclusion from the study.

12. Donated blood or plasma within 8 weeks before dose administration to a blood bank or blood donation center.

13. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 2 years before dose administration, or positive drug screening test reflecting consumption of illicit drugs.

14. History of alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 2 years before dose administration, or positive alcohol screen.

15. Known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen or hepatitis C antibodies, or have a positive result to the test for HIV antibodies at screening.

16. Smokes more than 10 cigarettes per day, or the equivalent in other tobacco products (self reported).

17. Part of the clinical site staff personnel or family members of the clinical site staff.

18. History of less than one to two bowel movements per day.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2014-10-08 (Actual); Study Completion 2014-10-08 (Actual)

PRIMARY OUTCOMES:
Total [14C]-radioactivity in biological matrices-Pharmacokinetics (PK) | Up to 12 days
  Biological matrices (whole blood, plasma, urine and feces) will be collected and analyzed for total [14C]-radioactivity
Cumulative excretion of total [14C]-radioactivity in urine and feces (PK) | Up to 12 days
  Urine and feces will be collected and analyzed for measurement of [14C]-radioactivity
Total [14C]-radioactivity whole blood-to-plasma ratios: PK | Up to 8 days
  Blood samples will be collected and analyzed for measurement of [14C]-radioactivity
Metabolite profiling/characterization in select biological matrices-PK | Up to 12 dyas
  Biological matrices (plasma, urine, and fecal samples) will be collected and select samples will undergo metabolite profiling/characterization
Peak (maximum) plasma concentration (Cmax) for total [14C]-radioactivity, [14C]-CC-122, and [14C]-metabolite(s), as appropriate PK | Up to 12 days
  Blood samples will be collected and analyzed; Maximum observed plasma or whole blood concentration for up to 168 hours postdose will be calculated and reported as appropriate
Area under the plasma concentration-time curve (AUC) for total [14C]-radioactivity, [14C]-CC-122, and [14C]-metabolite(s), as appropriate | Up to 12 days
  Blood samples will be collected and analyzed; Area under the concentration-time curve from time zero up to 168 hours postdose will be calculated and reported as appropriate
Time to maximum plasma concentration (Tmax) for total [14C]-radioactivity, [14C]-CC-122, and [14C]-metabolite(s), as appropriate | Up to 12 days
  Blood samples will be collected and analyzed; Time to reach the observed maximum (peak) concentration will be calculated and reported as appropriate.
Terminal elimination half-life (t1/2) for total [14C]-radioactivity, [14C]-CC-122, and [14C]-metabolite(s), as appropriate | Up to 12 days
  Blood samples will be collected and analyzed; Terminal half-life will be calculated and reported as appropriate

SECONDARY OUTCOMES:
The incidence, type, severity of adverse events (AE) | Up to 28 days following dose; AEs will be collected and recorded from the time the subjects signs Informed Consent throughthe 28 day period following the of last dose of study drug
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values regardless of etiology

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Mara, MD, Study Director — Celgene Corporation
Locations (1):
- Covance Clinical Research Unit Inc, Madison, Wisconsin, United States